CLINICAL TRIAL: NCT06656949
Title: A Prospective, Randomized Trial Comparing the Different Injection Sites of Indocyanine Green (ICG) in Sentinel Lymph Node Mapping in Patients With Endometrial Cancer
Brief Title: Sentinel Lymph Node Mapping With Different Injection Sites of ICG in Endometrium Cancer
Acronym: SLN-EC-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Youzhong Zhang, chief of OB&G department, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLL-202404-005-1
Record Dates: First submitted 2024-10-08; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: The study design is a two-arm, randomized, controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sentinel lymph node mapping with One injection site (cervix) group (Active Comparator): injecting indocyanine green (ICG) dye Intraoperative in cervix
  Interventions: Procedure: injecting indocyanine green (ICG) dye Intraoperative
- sentinel lymph node mapping with two injection site (cervix-uterus) group (Experimental): injecting indocyanine green (ICG) dye Intraoperative in cervix and uterus
  Interventions: Procedure: injecting indocyanine green (ICG) dye Intraoperative

INTERVENTIONS:
Procedure: injecting indocyanine green (ICG) dye Intraoperative — injecting indocyanine green (ICG) dye Intraoperative for patients with endometrial cancer

SUMMARY:
The primary goal of this prospective study is to define the efficacy of the sentinel lymph node biopsy (SLNB) procedure by comparing different method performed in patients with endometrial cancer. The aim of this study is to investigate whether the detection rate of sentinel lymph node (SLN) with two different injection sites may be increased compared to the standard use with single site (cervix) injection in endometrial cancer.

DETAILED DESCRIPTION:
The primary treatment for endometrial cancer involves total hysterectomy and bilateral salpingo-oophorectomy, with adjuvant radiotherapy and/or chemotherapy reserved for patients with advanced disease or who have risk factors for relapse. The tumor is confined to the uterus in 85% of endometrial cancers. Hence, it's controversial to perform systematic lymphadenectomy to all patients. The primary purpose of the present study is the to investigate the feasibility of sentinel lymph node determination in endometrial cancer patients operated via conventional laparoscopy. To determine sentinel lymph nodes cervical indocyanine green will be injected prior to the surgery. During the surgery using fluorescent imaging systems sentinel lymph nodes will be removed and examined by frozen section. Afterwards, systematic pelvic lymphadenectomy will be performed if sentinel lymph node is positive.

ELIGIBILITY:
Inclusion Criteria:

* • 1.Age >18 and <80 years old

  * 2. The pathological diagnosis was epithelial ovarian cancer
  * 3.Survival time is expected to exceed 3 months
  * 4.Signed consent form

Exclusion Criteria:

* 1. Patients with myocardial infarction or stroke, or unstable angina pectoris or decompensated heart function
* 2.Patients with a history of exhaustion or deep vein thrombosis;
* 3. Liver insufficiency (transaminase >2.5 times the upper limit of the standard);
* 4. Renal insufficiency (serum muscle liver >2 times the standard upper limit);
* 5. Pregnancy and perinatal patients;
* 6. History of major organ transplantation and immune disease;
* 7. Psychiatric condition or language barriers
* 8. Alcohol or drug abuser (current or previous)
* 9. Unable or unwilling to sign informed consent or comply with study requirements;
* 10. Patients with other malignant tumors.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
paraaortic Sentinel lymph node detection rates | intraoperative day0
  IGC positive Sentinel lymph node detection in paraaoritc lymph node will be assessed
Sentinel lymph node technique accuracy | postoperative up to day7
  Sensitivity and specificity measure of the sentinel lymph node for detecting the lymphatic metastasis

SECONDARY OUTCOMES:
Optimizing Sentinel lymph node detection procedure in endometrium cancer | intraoperative day 0
  Optimizing injectiong site, tow site injection vs one site injection
The difference Sentinel lymph node detection rate with Double Injection Sites and one injection site | intraoperative day 0
  assessing difference IGC positive sentinel lymph node detection rate with Double Injection Sites and one injection site
Postoperative complications | postoperative up to day 30
  Postoperative complications including damage of insestine , urethra and bladder

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital，Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No